CLINICAL TRIAL: NCT01810601
Title: Effect of Ultrasound Guided Embryo Transfer on Pregnancy Rates
Acronym: ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Noha Rabei, Assistent Professor, Obstet Gynecol, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: noharabei-1
Record Dates: First submitted 2013-03-12; First posted 2013-03-13 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Infertility
Keywords: Embryo transfer, transabdominal ultrasound, IVF, ICSI
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone; Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound guided embryo transfer (Experimental): GnRh, HMG, HCG, Progesterone 45 patients had ultrasound guided embryo transfer during ICSI
  Interventions: Drug: GnRh, HMG, HCG, Progesterone
- clinical touch technique (Placebo Comparator): GnRh, HMG, HCG, Progesterone 45 patients had embryo transfer using clinical touch technique during ICSI
  Interventions: Drug: GnRh, HMG, HCG, Progesterone

INTERVENTIONS:
Drug: GnRh, HMG, HCG, Progesterone — GnRh analogue (0.05 mg/day), HMG (150-300 iu/day), HCG (5000 iu/day), Progesterone (100 mg/day)

SUMMARY:
To assess the effect of transabdominal ultrasound guided embryo transfer on the pregnancy rates versus clinical touch technique

DETAILED DESCRIPTION:
A total of 90 patients undergoing treatment with ICSI were divided into 2 groups: group 1 (45 patients), had ultrasound guided embryo transfer and group 2 (45 patients), underwent embryo transfer using the clinical touch technique

ELIGIBILITY:
Inclusion Criteria:

* Age (20-39)
* Male factor infertility
* Ovarian factor infertility
* Unexplained infertility

Exclusion Criteria:

* Tubal factor infertility
* Endometriosis
* FSH > 16 iu/l on cycle day 3
* Less than 2 embryos grade A
* Difficult embryo transfer

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To assess clinical pregnancy rates after using ultrasound guided embryo transfer | After December, 2012

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R Ammar, MD, Study Director — Ain Shams University
Locations (1):
- IVF Unit, Ain Shams Maternity Hospital, Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Coroleu B, Barri PN, Carreras O, Belil I, Buxaderas R, Veiga A, Balasch J. Effect of using an echogenic catheter for ultrasound-guided embryo transfer in an IVF programme: a prospective, randomized, controlled study. Hum Reprod. 2006 Jul;21(7):1809-15. doi: 10.1093/humrep/del045. Epub 2006 Mar 23. PMID 16556674